CLINICAL TRIAL: NCT06028204
Title: The Role of the Lung Microbiome in Asthma and Its Influence on Treatment Response.
Brief Title: This is a 6-month Observational Study. Patients Included Will be Those Referred With a Possible Diagnosis or an Established Diagnosis of Asthma. It Will Look at the Association of the Asthma Microbiome and Disease Characteristics, Severity and Treatment Response.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: The Charitable Infirmary Charitable Trust (Unknown); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 23.29
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Biological Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Once all collected, the available samples will be processed for microbiome and host transcriptome profiling. Blood samples will be processed for complete blood count, immunoglobulin E and aeroallergen sensitivity. In addition blood will be processed for host immune profiling. Background control, oral rinse, nasopharyngeal swab, exhaled breath condensate, induced sputum and stool samples will be processed for microbiome. EBC and induced sputum will also be processed for host immune profiling. From the bronchoscopy cohort, all collected samples will undergo microbiome analysis. We will also perform host immune profiling on BAL samples. Endobronchial brushes will be processed for host transcriptome analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biologic Naïve Group: This will aim to include 50 patients who have been referred with possible asthma or have a diagnosis of asthma, and are established on treatment in the form of bronchodilators and/or inhaled corticosteroids who are not candidates for biologic therapy at present
- Biologic Group: This will aim to include 10 patients who have been referred with an established diagnosis of asthma and are on treatment in the form of bronchodilators and/or inhaled corticosteroids and have been selected as suitable candidates for commencing biologic therapy.
  Interventions: Drug: Biologic Agent

INTERVENTIONS:
Drug: Biologic Agent — Biologic group will have biological agent commenced if considered necessary as part of routine care.
  Groups: Biologic Group

SUMMARY:
The goal of this observational study is to investigate the role of the lung microbiome in patients with asthma and how it may influence the response to asthma specific treatments. This will be compared to patients who presented similarly but do not have a diagnosis of asthma.

The main aims are to:

1. Evaluate the influence of the microbiome on asthma phenotypes
2. Evaluate the influence of the microbiome on respiratory physiological change
3. Evaluate the effect of asthma treatment on the microbiome and the host response

Participants will be asked to provide a medical history focusing on their asthma and related co-morbidities such as sinus and reflux disease. They will have physiological parameters measured (spirometry, impulse oscillometry, fraction of exhaled nitric oxide). They will have samples collected to assess the upper and lower airway microbiome (oral rinse, nasopharyngeal swab, sputum, exhaled breath condensate and bronchoscopy) as well as the gut microbiome (stool). They will also have serum samples taken to perform host immune profiling (host transcriptome). They will be followed over six months observing how changes to asthma specific treatments, particularly inhaled corticosteroids and biologic agents can affect the microbiome

DETAILED DESCRIPTION:
VISIT 1 (Month 0) FACE TO FACE

* Once consented a study ID will be assigned, and basic demographic information taken.
* A standardized medical history will be taken to include target symptom history, exacerbation frequency and hospital admissions.
* A detailed co-morbid history will be taken as will a review of all previous asthma treatments. Validated symptom questionnaires will be completed during the study visits.
* All participants will be given an electronic PEFR monitor.
* Patients on or planned for inhaled therapy will be given an electronic adherence monitor.
* Pulmonary function testing will be performed including Spirometry, Impulse Oscillometry, Fraction of exhaled Nitric Oxide along with bronchodilator reversibility.
* Sample collection will include blood, oral rinse, nasopharyngeal swab, exhaled breath condensate, stool and induced sputum.
* A subset of patients will be consented for bronchoscopy for lower airway sampling.

VISIT 2,3, 4 (Month 1,2, 3) FACE TO FACE

* A detailed history of symptoms will be taken as will a review of all treatment changes.
* Validated symptom questionnaires will be completed during the study visits.
* PEFR and adherence device data from the previous month will be collected and new monitors and devices provided where needed.
* Pulmonary function testing will be performed as above.
* Sample collection will include blood, oral rinse, nasopharyngeal swab, EBC, stool and induced sputum as above.

VISIT 5 (Month 6) FACE TO FACE

* A detailed history of symptoms will be taken as will a review of all treatment changes. - Validated symptom questionnaires will be completed during the study visits.
* PEFR and adherence device data from the previous month will be collected and new monitors and devices provided where needed.
* Pulmonary function testing will be performed as above.
* Sample collection will include blood, oral rinse, nasopharyngeal swab, EBC, stool and induced sputum.
* A subset of patients who had bronchoscopy at VISIT 1 will have bronchoscopy performed again for corresponding sample collection.

PROCEDURES:

Questionnaires:

Validated symptom questionnaires will be completed during the study visits indicated previously. Asthma Control Test measures the adequacy of asthma control and change in asthma control which may occur spontaneously or in response to treatment. The GERD-Q and the SNOT-22 establish the presence and severity of co-morbid Gastro-oesophageal reflux disease and sinus disease, both common asthma co-morbidities, which may affect quality of life, symptom control and treatment response.

Investigations:

Pulmonary function testing will include spirometry, impulse oscillometry (IOS), Peak Expiratory Flow Rate (PEFR) measurement. Fraction of exhaled Nitric Oxide (FeNO), an established biomarker measured routinely in asthma clinics, will also be measured.

Bio-samples:

Background samples will be taken from sampling and storage equipment to examine for environmental contamination including sterile saline, nasopharyngeal swab, oral rinse/sputum pot container and the bronchoscope.

Blood tests will be drawn via phlebotomy and a single needle pass. The total quantity of blood volume drawn will be the minimally acceptable volume used in paediatric patients for research purposes. Maximum total sample volume is 50ml/10 teaspoons.

Oral samples will be collected using a standardized procedure in accordance with the Manual of Procedures for Human Microbiome Project. Study participants will rinse their mouth (swish/gargle) with 15 mL sterile normal saline for 1 min and will expectorate the contents of the mouth into a 50 mL centrifuge tube. Sample should be kept cold on ice until processing.

Nasopharyngeal swab will be collected inserted into each nostril for several seconds.

Induced sputum will be collected in selected patients using hypertonic saline where needed.

EBC will be collected using RTube where a one way breathing valve that allows contaminant free collection of 200 microlitres per minute in adults during normal breathing.

Stool will be collected in a sealable container and stored at -80 for further processing.

Bronchoscopy will be performed under moderate sedation with topical anaesthesia. A small camera is passed through the vocal cords into the upper then lower airways. For a bronchoalveolar lavage (BAL) a total of 60ml of normal saline will be instilled into a pulmonary lobe and the return will be collected for analysis. An endothelial brushing (EB) involves the introduction of a small brush via the bronchoscope to gently brush the airway walls to collect epithelial cells for analysis for morphological and functional studies.

SAMPLE PROCESSING:

Samples will be processed and stored in RCSI. Once all collected, the available samples will be transferred to New York University Hospitals (for our collaborator Dr. Leopoldo Segal), to be processed for microbiome and host transcriptome profiling.

Blood samples will be processed for complete blood count, immunoglobulin E and aeroallergen sensitivity. In addition blood will be processed for host immune profiling.

Background control, oral rinse, nasopharyngeal swab, EBC, induced sputum and stool samples will be processed for microbiome. EBC and induced sputum will also be processed for host immune profiling.

From the bronchoscopy cohort, all collected samples will undergo microbiome analysis. We will also perform host immune profiling on BAL samples. Endobronchial brushes will be processed for host transcriptome analysis.

* Host immune profiling: Cytokine analysis of samples will be done by Luminex multiplex
* 16S rRNA gene sequencing (microbiome): Nucleic acid extraction, 16S rRNA gene amplification, and purification will be performed and sequencing will be performed on a MiSeq platform (Illumina). This data will be analysed with Quantitative Insights Into Microbial Ecology (QIIME).
* Bulk RNAseq (host transciptome): RNAseq will be performed on bronchial epithelial cells obtained by bronchial brushing (EB), using the Hi-seq /Illumina platform. Sequences will be aligned against the hg19 ensemble reference genome, subsequent gene counting will be performed using featureCounts and differential gene expression will be calculated using the DESeq2 package with an adjusted p-value <0.05. Ingenuity Pathway Analysis (IPA) will used to identify top biological functions. Genes will be mapped to Ensembl IDs and subsequently to KEGG pathways. We will also use analytical approaches designed to establish an immunological profiling such as CIBERSORT.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Patients able to give informed consent
* Patients who have been referred with possible asthma or have an established diagnosis of asthma

Exclusion Criteria:

* Patients <18 years
* Patients unable to give informed consent
* Patients who are or intend to become pregnant during the study period
* Other co-existent respiratory diagnosis e.g. bronchiectasis, COPD, Pulmonary fibrosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient referred with a possible diagnosis of asthma or established diagnosis of asthma to hospital or the Respiratory Outpatient Department
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Describe microbiome signature across the spectrum of asthma severity | 2 years
  We expect an increasingly dysbiotic signature in the respiratory microbiome of patients with severe asthma.
Establish if there is any association between asthma phenotype and microbiome signature | 2 years
  We expect to see a correlation between dysbiosis in the respiratory microbiome and changes in symptom control and physiological parameters.
Determine whether microbiome signature can predict treatment response or resistence | 2 years
  We expect to identify a microbial signature in the respiratory microbiome associated with treatment response, to both biological therapy as well as inhaled corticosteroids.

IPD SHARING:
Plan to Share IPD: Undecided
If coded data were to be used again, further patient consent, ethical and data protection approval would be required.